CLINICAL TRIAL: NCT05776901
Title: Mobile Health (mHealth) Application Called CBCT Sessions to Treat and Reduce Elevated Stress Among Students (C-STRESS)
Brief Title: C-STRESS: A Mental Health App for College Students With Depression
Acronym: C-STRESS
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Grant termination without continuation.
Sponsor: Benten Technologies, Inc. (Industry)
Collaborators: University of California, Irvine (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Tony Ma, President, Benten Technologies, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: C-STRESS; R44MH121219 (NIH)
Record Dates: First submitted 2023-02-28; First posted 2023-03-20 (Actual); Results first posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Depression; Anxiety; Stress, Psychological; Mobile Phone Use
Keywords: Depression; Anxiety; Stress; mHealth; college students
MeSH Terms: conditions — Depression; Anxiety Disorders; Stress, Psychological; Cell Phone Use

STUDY DESIGN:
Intervention Model Description: All participants enrolled in the study were asked to use the C-STRESS app daily for 6 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: C-STRESS — Participants were asked to use the C-STRESS app daily for 6 weeks to participate in Cognitively Based Compassion Training (CBCT) lessons, watch guided meditation videos, complete short reflective exercises, and engage with other content provided in C-STRESS (i.e., attending drop-in sessions, journaling, completing mood and wellbeing check-ins, and reading educational articles on depression, anxiety, and stress)

SUMMARY:
The goal of this pilot study is to examine the feasibility of the prototype C-STRESS app with 3 college students from UCI with clinically significant depression (scored ≥ 10 on the Patient Health Questionnaire-9). The main question it aims to answer is: whether the prototype C-STRESS is useful for college students to manage daily stress and depression symptoms.

Participants were asked to use the C-STRESS app daily for 6 weeks to participate in CBCT lessons, watch guided meditation videos, complete short reflective exercises, and engage with other content provided in C-STRESS (i.e., attending drop-in sessions, journaling, completing mood and wellbeing check-ins, and reading educational articles on depression, anxiety, and stress). At the end of week 3 and 6, participants completed 6 online surveys (System Usability Scale, Technology Acceptance Model, Patient Health Questionnaire-9, General Anxiety Disorder-7, Health Related Quality of Life-4, and Brief-COPE) to assess C-STRESS's usability/feasibility and changes in depressive symptoms and coping styles over the study period.

DETAILED DESCRIPTION:
More than half of U.S. college students experience significant symptoms of depression, anxiety or stress, and three-fourths of these college students do not obtain professional help due to overburdened mental health services at universities and colleges. Prevalence of mental disorders and inadequate utilization of mental health services is a particularly severe problem for minority students and community college students. Cognitively Based Compassion Training (CBCT) has been administered to a variety of populations, including college students (undergraduate students, medical school students) and younger adolescents in prior completed studies, that collectively showed that CBCT can significantly strengthen cognitive resilience to stress and substantially reduce depressive symptoms, stress-associated systemic inflammation, improve emotional regulation (including impulse control) and mindfulness; increase compassion, and improve empathetic accuracy (measured by fMRI) - a critical skill that aims at cultivating relationships and connection to others. Currently, as a face-to-face program, CBCT certification at Emory takes 1 year to complete, and there are only 48 CBCT instructors. Due to the course duration, location, and time-intensive requirement for certification, CBCT has limited reach and scalability in its current instructional model despite growing demands.

The research team developed C-STRESS, a digital treatment intervention that leverages CBCT to improve the mental health of college students. C-STRESS adapts the traditional intervention modality (face-to-face) of CBCT in the form of micro-learning and provides personalization options including virtual companions and an animated visual cue of growing a garden to promote student engagement. Using co-design sessions with college students, the research team developed other features in C-STRESS to address the target population's needs when it comes to using a mobile app for mental health care, including an audiovisual library of guided meditation and resources, journaling, virtual drop-ins with CBCT instructors, mood and wellbeing tracking, and crisis helpline.

The research team recruited an independent convenience sample of 3 UCI undergraduate and graduate students to pilot test the initial content (introduction and modules 0-3) of the prototype C-STRESS mobile application. Participants completed measures via REDCap. Once enrolled, participants met with a member of the research team via Zoom to a) download the prototype app, b) complete app orientation (eg. indicate reason(s) for using the app, indicate color scheme & frequency of notification preferences, select avatar if desired, etc.), c) begin to explore the app and its functionality with a research team member available to provide technical assistance, and d) complete the System Usability Scale and Technology Acceptance Model questionnaires via REDCap survey link. After the app orientation, participants were asked to use the prototype C-STRESS application at least once per day for 6 weeks. Daily usage ranged from approximately 2 minutes (opening the app and performing a one-minute meditation) to as much time as the participant desires (opening the app, completing available content, and unlimited meditation/reflection/journaling, etc. multiple times per day). At the end of week 3 (timepoint 1) and week 6 (timepoint 2), the participants were asked to complete measures via REDCap survey to assess C-STRESS's usability/feasibility and changes in depressive symptoms and coping styles over the 6-week study period.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate or graduate students
* Enrolled at University of California Irvine (UCI)
* Between the ages of 18-30
* Speak and understand English
* Have access to the internet for 6 weeks to participate in study activities via Zoom
* Report clinically significant depression (scores ≥ 10 on the Patient Health Questionnaire-9)
* Have a smart phone with either iPhone Operating System (iOS) or android operating system

Exclusion Criteria:

* Report active suicidal ideation unless they obtain a written note of approval from a psychiatric provider
* Female student who self-report pregnancy or plans to become pregnant within the next 3 months

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2022-05-04 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UCI, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited via print, email, or electronic posting of flyer on UCI websites or affiliated social media and locations in and around UCI campus from March 16 to May 31, 2022. All three participants were enrolled on May 04, 2022. Due to grant termination, final collection of data for the primary outcome was on May 25, 2022, which allowed us to collect data at baseline and week 3, but not perform data collection at week 6 due to grant termination.
Pre-assignment Details: All participants were assigned to the C-STRESS arm. Participants who reported active suicidal ideation and female students who self-reported pregnant or plans to become pregnant within the next 3 months were excluded.
Period: Overall Study
Arm/Group | C-STRESS
Started (Milestone 1 (Week 1): Completion of the C-STRESS app orientation session and the SUS questionnaire at the baseline.) | 3
Week 3 (Milestone 2 (Week 3): Completion of the SUS questionnaire at week 3) | 3
Week 6 (Milestone 3: Completion of the SUS questionnaire at week 6. The collection of data was not completed due to grant termination.) | 0
Completed | 0
Not Completed | 3
Not completed — Covid delays and grant termination without continuation. | 3

BASELINE CHARACTERISTICS:
Groups:
- C-STRESS: Participants were asked to use the C-STRESS app daily for 6 weeks to participate in CBCT lessons, watch guided meditation videos, complete short reflective exercises, and engage with other content provided in C-STRESS (i.e., attending drop-in sessions, journaling, completing mood and wellbeing check-ins, and reading educational articles on depression, anxiety, and stress)
Arm/Group | C-STRESS
Number analyzed (Participants) | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.67 (1.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 1
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3
System Usability Scale [Mean (Standard Deviation); unit: score on a scale] — The System Usability Scale (SUS) is a reliable assessment tool for evaluating the perceived usability and ease of use of a product or service. The scale comprises ten questions, each with five possible responses, ranging from 1 (Strongly disagree) to 5 (Strongly agree). The participant's response to each question is converted to a score, added together and then multiplied by 2.5 to convert their original responses to a score of 0-100. A higher score indicates higher perceived usability and ease of use of a product or service.
  score on a scale | 54.58 (20.59)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline System Usability Scale Scores at Week 3 and Week 6
Description: The System Usability Scale (SUS) is a reliable assessment tool for evaluating the perceived usability and ease of use of a product or service. The scale comprises ten questions, each with five possible responses, ranging from 1 (Strongly disagree) to 5 (Strongly agree). The participant's response to each question is converted to a score, added together and then multiplied by 2.5 to convert their original responses to a score of 0-100. A higher score indicates higher perceived usability and ease of use of a product or service. SUS was assessed at both the baseline and week 3. However, there was no assessment of SUS in week 6 due to grant termination.
Time Frame: Baseline, week 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | C-STRESS
Number analyzed (Participants) | 3
score on a scale
  Milestone 1 (week 1): Completion of the C-STRESS app orientation session and the SUS questionnaire | 71.67 (11.61)
  Milestone 2: Completion of the SUS questionnaire at week 3 | 37.5 (11.37)
  Change from baseline SUS scores at week 3 | 34.17 (20.45)
Statistical Analysis 1: Comparison: C-STRESS; Test type: Other — Descriptive statistics and measures of central tendency, including mean, median, and standard deviation of the System Usability Scores collected from the baseline and week 3 were computed. Then, a two-sided, paired sample t-test was conducted to evaluate the change in mean System Usability Scores from baseline at week 3; p < 0.05, t-test, 2 sided; Mean diff in SUS from baseline at week 3 = 34.17, 95% CI 2-sided [-28.04 to 96.37], Standard Error of Mean 14.49

ADVERSE EVENTS:
Time Frame: Adverse event data for the entire study were collected over 27 days, starting from the enrollment of the first participant on May 04, 2022, to May 31, 2022. Adverse event data for each participant were collected twice over 3 weeks, at the baseline and 3-week follow-up.
Description: Adverse event data for each participant were assessed at the baseline and 3-week follow-up using the Patient Health Questionnaire 9 to evaluate their risk for suicide ideation and self-harm.
Arm/Group | C-STRESS
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

LIMITATIONS AND CAVEATS:
The enrollment of only 3 female participants compromised the generalizability of this study in two ways. Firstly, with such a small sample size, it is challenging to draw broad conclusions regarding the usability of the C-STRESS app for the boarder population.

Secondly, having an imbalanced representation of gender can limit the ability to detect potential gender-specific effects or gender differences.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-03-16): https://cdn.clinicaltrials.gov/large-docs/01/NCT05776901/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-09): https://cdn.clinicaltrials.gov/large-docs/01/NCT05776901/SAP_001.pdf